CLINICAL TRIAL: NCT01203982
Title: Effect of Intensive Lipid Lowering Treatment Compared to Moderate Lipid Lowering Treatment on Carotid Intima Media Thickness and Its Relation to Plaque Components of the Coronary Arteries in Patients With ST-Segment Elevation Acute Myocardial Infarction
Brief Title: Effect of Intensive Lipid Lowering Treatment Compared to Moderate Lipid Lowering Treatment on Carotid Intima-media Thickness (CIMT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Rasmus Egede, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VF-20060060
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: ST-segment Elevation Myocardial Infarction; Subclinical Carotid Atherosclerosis
Keywords: CIMT; IVUS-VH; Coronary artery disease
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Coronary Artery Disease | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin 5mg (Active Comparator): Rosuvastatin 5mg/day
  Interventions: Drug: Rosuvastatin
- Rosuvastatin 40mg (Active Comparator): Rosuvastatin 40mg/day
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 5mg/day for one year
  Other Names: Crestor
  Arms: Rosuvastatin 5mg
Drug: Rosuvastatin — Rosuvastatin 40mg/day for one year
  Other Names: Crestor
  Arms: Rosuvastatin 40mg

SUMMARY:
The aim of this study was to measure the effect of moderate and intensive lipid-lowering treatment with rosuvastatin on the carotid intima-media thickness (CIMT) as a surrogate marker of cardiovascular risk.

DETAILED DESCRIPTION:
The aim of this study was to measure the effect of moderate (5mg) and intensive (40mg) lipid-lowering treatment with rosuvastatin on the carotid intima-media thickness as a surrogate marker of cardiovascular risk and to obtain whether CIMT correlated with the plaque components in coronary arteries evaluated with Intravascular Ultrasound Virtual Histology (IVUS-VH).

ELIGIBILITY:
Inclusion Criteria:

1. STEMI,
2. no prior treatment with statins and
3. a non significant lesion in one of the two non-culprit coronary arteries. -

Exclusion Criteria:

1. age below 18 or above 81 years,
2. unconscious patients,
3. serum creatinine > 176μmol/L,
4. total-cholesterol > 7.0 mmol/l,
5. hypothyroidism ((TSH > 1.5 x ULN (upper limit of normal)),
6. current liver disease (ALAT > 2 x ULN),
7. unexplained creatine kinase > 3 x ULN,
8. alcohol or drug abuse within the last five years,
9. prior myopathy or serious hypersensitivity reaction caused by statins,
10. women with childbearing potential who were not using chemical or mechanical contraception,
11. pregnant or breastfeeding women,
12. history of malignancy unless a disease-free period of more than five years was present,
13. patients with abnormal lung function test (LFT),
14. participation in another investigational drug study less than four weeks before enrolment in the present study,
15. treatment with cyclosporine or fibrates. -

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-11; Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
change from baseline in mean CIMT | baseline, 6month, 12 month
  Average of the far wall of common and bulbus carotid artery

SECONDARY OUTCOMES:
changes from baseline in max CIMT | baseline, 6month, 12 month
change from baseline in mean common CIMT | baaseline, 6month 12 month
change from baseline in max common CIMT | baseline, 6month 12month
change from baseline in mean bulbus CIMT | Baseline, 6month 12 month
change from baseline in max bulbus CIMT | baseline, 6month 12month
change from baseline in lipid values | baseline, 6month 12month
correlation between CIMT measurements and lipid values | Baseline, 6month 12 month
correlation between CIMT measurements and plaque components evaluated by IVUS-VH | Baseline, 6month 12month

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Odense University Hospital, Odense, Fuenen, Denmark